CLINICAL TRIAL: NCT03460600
Title: OCT Documents Vitreo-papillary Traction
Brief Title: Vitreo-papillary Traction as an Entity Identified by Optical Coherence Tomography (OCT).
Status: Completed | Type: Observational
Sponsor: Dr. S.S. Michel Clinic (Other)
Responsible Party: Principal Investigator, Dr. Shawkat Michel, ophthalmologist, Dr. S.S. Michel Clinic
Other Study IDs: vitreo-papillary traction
Record Dates: First submitted 2018-02-28; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Tomography, Optical Coherence
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Optical Coherence Tomography (OCT) — Optical Coherence Tomography is a fairly new imaging technique in ophthalmology

SUMMARY:
Optical Coherence Tomography (OCT) is a relatively new imaging technique in ophthalmology. This clear and documented imaging identified new diseases/ observations that were not previously known.

DETAILED DESCRIPTION:
In ophthalmology vitreo-macular adhesion, vitreo-macular traction and posterior vitreous detachment were recognized entities for a long time. On the other hand vitreo-papillary adhesion/ traction is a fairly new concept in ophthalmology that became known after the use of OCT in ophthalmology imaging. Reasons, effects and ways of treatment of vitreo-papillary traction will take some time to evolve. The case study in which this traction was documented was initiated by an observation of a persistent, tiny single retinal hemorrhage above the optic disc of an eye. The patient was completely asymptomatic because of the vitreo-papillary traction but the OCT documentation of the case was so clear and striking.

ELIGIBILITY:
Inclusion Criteria:

* any human subject that is found to have VPT by OCT.

Exclusion Criteria:

-

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any himan subject that is found to have VPT by OCT.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Tomography, Optical Coherence (OCT) | through study completion, usually one day.
  Vitreo-papillary traction (VPT) is a relatively new finding in ophthalmology that became very well known and documented by Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: shawkat michel, Principal Investigator — Dr. S.S. Michel Clinic Edmonton, Alberta Canada
Locations (1):
- Dr. S.S. Michel Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
if someone is interested in this case he/ she needs to send a new/ previously unused USB and I will transfer OCT images available to him/ her.
Supporting Information: CSR
Time Frame: starting now for three months till May 31, 2018.
Access Criteria: send a new USB and a postage paid return envelop.